CLINICAL TRIAL: NCT02386930
Title: Behavioral Lifestyle Intervention Study (BLIS) in Patients With Type 2 Diabetes in UAE: A Randomized Controlled Trial in Real Life Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rashid Centre for Diabetes and Research (Other)
Responsible Party: Principal Investigator, Sarah Qassim Abdi, Clinical dietitian, Rashid Centre for Diabetes and Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 032013-07
Record Dates: First submitted 2015-03-07; First posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: Cognitive behavior therapy; Lifestyle modification; HbA1c; Carbohydrates
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavrioal Lifestyle modification (Experimental)
  Interventions: Behavioral: Behvarioal lifestyle modification
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Behvarioal lifestyle modification — A six months behavioral lifestyle program composed of 8 sessions; 4 individual consultations and 4 telephonic calls. The cognitive behavior theory (CBT) is the underpinning theory for the lifestyle intervention; hence CBT behavioral strategies like self monitoring and goal setting are used to improve compliance to healthy lifestyle practices
  Arms: Behavrioal Lifestyle modification

SUMMARY:
The primary purpose of this study is to develop a behavioral lifestyle intervention and evaluate its effectiveness in improving the glycemic control in patients with type 2 diabetes in real life setting. This is because ambiguity still exists on the effectiveness of behavioral lifestyle interventions in routine clinical practice despite of the efficacy of large randomized controlled trials, suggesting the need for more research in this area.

ELIGIBILITY:
Inclusion Criteria:

Females or males. Type 2 diabetes. BMI (kg/ m²) ≥ 25. Age 18-60 years old. HbA1c > 7%.

Exclusion Criteria:

major physical activity disability that restricts participation in moderate physical activity.

serious heart condition like heart failure, heart attack, stroke within the last 3 months.

participating in a weight management or lifestyle program. presence of proliferative retinopathy or kidney failure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
HbA1c% | 6 months

SECONDARY OUTCOMES:
Weight | 6 months
Body composition analysis | 6 months
Lipid profile ( serum cholesterol, LDL, HDL, triglycerides) | 6 months
Blood presssure (systolic and diastolic) | 6 months
carbohydrates intake in grams | 6 months
physical exercise in minutes per day | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rashid Centre for Diabetes and Research, Ajman, United Arab Emirates